CLINICAL TRIAL: NCT05125302
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Single-attack Study to Evaluate the Efficacy, Safety, Tolerability, and Pharmacokinetics of Oral Ubrogepant in the Acute Treatment of Migraine With or Without Aura in Children and Adolescents (Ages 6-17)
Brief Title: Study to Assess Adverse Events and Disease Activity of Oral Ubrogepant Tablets for the Acute Treatment of Migraine in Children and Adolescents (Ages 6-17)
Acronym: Ubro Peds
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3110-305-002
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Migraine
Keywords: Migraine; Ubrogepant; Ubrelvy; PERISCOPE
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- PK Cohort: Ubrogepant Dose A (Experimental): Participants aged 6 to 11 will receive oral tablets of ubrogepant for PK analysis to determine appropriate dose for main study.
  Interventions: Drug: Ubrogepant
- PK Cohort: Ubrogepant Dose B (Experimental): Participants aged 6 to 11 will receive oral tablets of ubrogepant for PK analysis to determine appropriate dose for main study.
  Interventions: Drug: Ubrogepant
- Main Study: Children Ubrogepant Low Dose (Experimental): Participants aged 6 to 11 (after dose selection) will receive oral tablets of low dose ubrogepant for qualifying migraine attack. Participants have the option to take a second dose of ubrogepant or rescue medication, starting 2 hours after initial dose for headache of moderate/severe intensity.
  Interventions: Drug: Ubrogepant
- Main Study: Children Ubrogepant High Dose (Experimental): Participants aged 6 to 11 (after dose selection) will receive oral tablets of high dose ubrogepant Dose B for qualifying migraine attack. Participants have the option to take a second dose of ubrogepant or rescue medication, starting 2 hours after initial dose for headache of moderate/severe intensity.
  Interventions: Drug: Ubrogepant
- Main Study: Children Ubrogepant Placebo (Placebo Comparator): Participants aged 6 to 11 (after dose selection) will receive oral tablets of placebo-matching ubrogepant for qualifying migraine attack. Participants have the option to take a second dose of placebo-matching ubrogepant or rescue medication, starting 2 hours after initial dose for headache of moderate/severe intensity.
  Interventions: Drug: Placebo-Matching Ubrogepant
- Main Study: Adolescents Ubrogepant Low Dose (Experimental): Participants aged 12 to 17 will receive oral tablets of ubrogepant low dose for qualifying migraine attack. Participants have the option to take a second dose of ubrogepant or rescue medication, starting 2 hours after initial dose for headache of moderate/severe intensity.
  Interventions: Drug: Ubrogepant
- Main Study: Adolescents Ubrogepant High Dose (Experimental): Participants aged 12 to 17 will receive oral tablets of ubrogepant high dose or qualifying migraine attack. Participants have the option to take a second dose of ubrogepant or rescue medication, starting 2 hours after initial dose for headache of moderate/severe intensity.
  Interventions: Drug: Ubrogepant
- Main Study: Adolescents Ubrogepant Placebo (Placebo Comparator): Participants aged 12 to 17 will receive oral tablets of placebo-matching ubrogepant for qualifying migraine attack. Participants have the option to take a second dose of placebo-matching ubrogepant or rescue medication, starting 2 hours after initial dose for headache of moderate/severe intensity.
  Interventions: Drug: Placebo-Matching Ubrogepant

INTERVENTIONS:
Drug: Ubrogepant — Oral Tablet
  Other Names: Ubrelvy
  Arms: Main Study: Adolescents Ubrogepant High Dose; Main Study: Adolescents Ubrogepant Low Dose; Main Study: Children Ubrogepant High Dose; Main Study: Children Ubrogepant Low Dose; PK Cohort: Ubrogepant Dose A; PK Cohort: Ubrogepant Dose B
Drug: Placebo-Matching Ubrogepant — Oral Tablet
  Arms: Main Study: Adolescents Ubrogepant Placebo; Main Study: Children Ubrogepant Placebo

SUMMARY:
Migraine is a common neurological disorder typically characterized by attacks of throbbing, moderate to severe headache, often associated with nausea, vomiting, and sensitivity to light and sound. Migraine is extremely common and disabling in children. The purpose of this study is to evaluate how safe and effective ubrogepant is in the acute treatment of migraine in children and adolescents.

Ubrogepant is a drug approved for the acute treatment of migraine in adults. Children and adolescents (aged 6-17 years) with a history of migraine will be enrolled. The study will include 2 cohorts of participants - PK Cohort and Main Study (non-PK cohort). Participants aged 6-11 years in the PK Cohort will receive Dose A or Dose B of Ubrogepant for PK analysis to determine dose selection for the main study. In the main study, after dose selection, children aged 6-11 years will be randomized to receive either low or high dose of Ubrogepant or placebo. There is a 1 in 3 chance that a participant will be assigned to placebo. Adolescents aged 12-17 years will be randomized to receive either low or high dose of Ubrogepant or placebo with a 1 in 3 chance of placebo assignment.

For qualifying migraine attacks, participants will receive oral tablets of the double-blind study intervention. There will be an option to take a second dose of double-blind study intervention (identical to initial dose), or rescue medication, at least 2 hours after the initial dose, for headache of moderate/severe intensity. Around 1059 participants will be enrolled in the study in approximately 120 sites in the United States. The study duration will be up to 6 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* A history of migraine with or without aura consistent with a diagnosis according to the International Classification of Headache Disorders (ICHD-3) for at least 6 months.
* By history, the participant's migraines typically last between 3 and 72 hours if untreated or treated unsuccessfully and migraine episodes are separated by at least 48 hours of headache pain freedom.
* History of 1 to 14 migraine attacks per month with moderate to severe headache in each of the 2 months prior to screening (Visit 1).
* Current or past use of at least 1 oral medication (over-the-counter medication or prescription medication) for the acute treatment of migraine.
* For main study participants, treatment of a qualifying migraine with single-blind placebo during the screening period and completion of 2-hour headache pain assessment.
* Weight is ≥ 20 kg (44 pounds) and < 135 kg (298 pounds)
* Per investigator judgment, participant is able to swallow or can learn to swallow study intervention.
* The participant is able to understand and complete the study questionnaires and eDiary. Participants who need assistance with reading the assessments may be assisted by a parent or guardian.

Exclusion Criteria:

* Any clinically significant hematologic, endocrine, pulmonary, renal, hepatic, gastrointestinal, cardiovascular or neurologic disease.
* In the opinion of the investigator, other confounding pain syndromes, confounding psychiatric conditions, or other significant neurological disorders other than migraine.
* History of malignancy in the 5 years prior to Visit 1.
* History of any prior gastrointestinal conditions (eg, diarrhea syndromes, inflammatory bowel disease) that may affect the absorption or metabolism of the study intervention.
* Significant risk of self-harm, based on clinical interview and responses on the Columbia-Suicide Severity Rating Scale (C-SSRS), or of harm to others; participants must be excluded if they report suicidal ideation with intent, with or without a plan, (ie, Type 4 or 5 on the C-SSRS) in the past 6 months or report suicidal behavior in the last 6 months prior to Visit 1 or Visit 2 assessments.
* At Visit 1, current alcohol or drug abuse or dependence per investigator's judgment.
* For main study participants, no headache at the 2-hour post dose assessment after taking single-blind placebo for a qualifying migraine during screening period (ie, placebo responder).
* A current diagnosis of chronic migraine as defined by ICHD-3
* Participants who overuse medication for migraine defined as use of opioids or barbiturates > 2 days/month, triptans or ergots ≥ 10 days/month, simple analgesics (eg, aspirin, NSAIDs, acetaminophen) ≥ 15 days/month or any combination of triptans, ergots, or simple analgesics (eg, aspirin, NSAIDs, acetaminophen) ≥ 10 days/month in the 3 months prior to Visit 1 per investigator's judgment.
* Difficulty distinguishing migraine headache from tension-type or other headaches.
* Has a history of migraine aura with diplopia or impairment of level of consciousness, hemiplegic migraine, or retinal migraine as defined by ICHD-3.
* Has a current diagnosis of new persistent daily headache, trigeminal autonomic cephalgia (eg, cluster headache), or painful cranial neuropathy as defined by ICHD-3
* Required in-hospital (excluding emergency department visits) treatment for migraines 3 or more times in the 6 months prior to Visit 1.
* Requirement for any medication (eg, barbiturates) or diet (eg, grapefruit juice) that is on the list of prohibited concomitant medications that cannot be discontinued or switched to an allowable, alternative medication at Visit 1.
* Previous exposure, within the last 6 months, to injectable monoclonal antibodies blocking the calcitonin gene-related peptide (CGRP) pathway
* History of hypersensitivity or clinically significant adverse reaction to a CGRP receptor antagonist or hypersensitivity to any component of the study interventions, ubrogepant or placebo.
* Currently participating or has participated in a study with an investigational compound or device within 30 days prior to Visit 1

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1059 (Estimated)
Dates: Start 2022-01-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with Pain Freedom at 2 Hours After the Initial Dose in pediatric participants aged 6 to 17 years | 2 hours after initial dose
  Pain Freedom is defined as a reduction in headache severity from moderate/severe at baseline to no pain.

SECONDARY OUTCOMES:
Percentage of participants with Pain Freedom at 2 Hours After the Initial Dose in pediatric participants aged 12 to 17 years | 2 hours after initial dose
  Pain Freedom is defined as a reduction in headache severity from moderate/severe at baseline to
Percentage of participants with Pain Relief at 2 Hours After the Initial Dose in pediatric participants aged 12 to 17 years | 2 hours after initial dose
  Pain Relief is defined as a reduction in headache severity from moderate/severe at baseline to mild or no pain.
Percentage of Participants With Sustained Pain Freedom From 2 to 24 Hours After Initial Dose in pediatric participants aged 6 to 17 years | 2 to 24 hours after initial dose
  Sustained pain freedom was defined as a pain freedom at 2 hours with no administration of either rescue medication or the second dose of study drug, and with no occurrence thereafter of a mild/moderate/severe headache up to 24 hours after dosing with study drug.
Percentage of participants that used rescue medication (including a second dose of study intervention) within 24 hours after the initial dose in pediatric participants aged 6 to 17 years | 24 hours after initial dose
Percentage of Participants With Absence of the Most Bothersome Migraine-Associated Symptom Identified at Baseline at 2-Hours After Initial Dose in pediatric participants aged 6 to 17 years | Baseline (Predose) to 2 hours after initial dose
  The most bothersome migraine-associated symptom was the symptom (photophobia, phonophobia or nausea) present at pre-dose baseline identified by the participant to be 'most bothersome'.
Percentage of Participants With Absence of the Most Bothersome Migraine-Associated Symptom Identified at Baseline at 2-Hours After Initial Dose in pediatric participants aged 12 to 17 years | Baseline (Predose) to 2 hours after initial dose
  The most bothersome migraine-associated symptom was the symptom (photophobia, phonophobia or nausea) present at pre-dose baseline identified by the participant to be 'most bothersome'.
Percentage of participants with Pain Freedom at 2 Hours After the Initial Dose in pediatric participants aged 6 to 11 years | 2 hours after initial dose
  Pain Freedom is defined as a reduction in headache severity from moderate/severe at baseline to no pain.
Percentage of Participants With the Absence of Photophobia at 2 Hours After the Initial Dose in pediatric participants aged 6 to 17 years | 2 hours after initial dose
  Photophobia was defined as sensitivity to light, a migraine-associated symptom.
Percentage of Participants With the Absence of Phonophobia at 2 Hours After the Initial Dose in pediatric participants aged 6 to 17 years | 2 hours after initial dose
  Phonophobia was defined as sensitivity to sound, a migraine-associated symptom.
Percentage of Participants With the Absence of Nausea at 2 Hours After the Initial Dose in pediatric participants aged 6 to 17 years | 2 hours after initial dose
  Nausea was a migraine-associated symptom.
Number of Participants with Adverse Events (AE) | Up to 6 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of Participants with Abnormal Change in Clinical Laboratory Test Results Like Hematology will be Assessed in pediatric participants aged 6 to 17 years | Up to 6 months
  Percentage of participants with abnormal change in clinical laboratory test results like hematology will be assessed.
Change From Baseline in Electrocardiograms (ECGs) in pediatric participants aged 6 to 17 years | Up to 6 months
  12-lead resting ECGs will be recorded. Parameters include heart rate, PR interval, QT interval, QRS duration, and QT interval corrected using Fridericia's formula (QTcF).
Percentage of Participants with Abnormal Change From Baseline in Vital Sign Measurements in pediatric participants aged 6 to 17 years | Up to 6 months
  Percentage of participants with abnormal change from baseline in vital sign measurements like systolic and diastolic blood pressure will be assessed.
Percentage of patients with suicidal ideation or suicidal behavior | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (122):
- United States (118):
  - Rehabilitation & Neurological Services /ID# 229969, Huntsville, Alabama
  - The Center for Clinical Trials - Saraland /ID# 231546, Saraland, Alabama
  - Velocity Clinical Research - Phoenix /ID# 274478, Phoenix, Arizona
  - HealthStar Research Glenwood /ID# 275303, Glenwood, Arkansas
  - HealthStar Research of Hot Springs PLLC /ID# 273256, Hot Springs, Arkansas
  - Preferred Research Partners /ID# 230725, Little Rock, Arkansas
  - Advanced Research Center /ID# 227962, Anaheim, California
  - Neuro Pain Research Center /ID# 227966, Fresno, California
  - Alliance for Research Alliance for Wellness /ID# 230546, Long Beach, California
  - Children's Hospital Los Angeles /ID# 230596, Los Angeles, California
  - Excell Research, Inc /ID# 230899, Oceanside, California
  - Paradigm Clinical Research - San Diego /ID# 269608, San Diego, California
  - Lumos Clinical Research Center /ID# 231267, San Jose, California
  - Pacific Clinical Research Management Group /ID# 231636, Upland, California
  - Sunwise Clinical Research /ID# 230971, Walnut Creek, California
  - Amicis Research Center /ID# 272621, Winnetka, California
  - Children's Hospital Colorado - Aurora /ID# 231879, Aurora, Colorado
  - IMMUNOe Research Centers /ID# 230879, Centennial, Colorado
  - MCB Clinical Research Centers /ID# 231625, Colorado Springs, Colorado
  - New England Institute for Clinical Research /ID# 230635, Stamford, Connecticut
  - Emerson Clinical Research Inst /ID# 231693, Washington D.C., District of Columbia
  - Encore Medical Research of Boynton Beach LLC /ID# 246833, Boynton Beach, Florida
  - Gulf Coast Clinical Research Center /ID# 230020, Fort Myers, Florida
  - Sarkis Clinical Trials /ID# 227956, Gainesville, Florida
  - Northwest Florida Clinical Research Group, LLC /ID# 231069, Gulf Breeze, Florida
  - AGA Clinical Trials /ID# 230554, Hialeah, Florida
  - Encore Medical Research /ID# 245682, Hollywood, Florida
  - Advanced Research Institute of Miami /ID# 230292, Homestead, Florida
  - Auzmer Research /ID# 239251, Lakeland, Florida
  - Columbus Clinical Services, Llc /Id# 230880, Miami, Florida
  - My Preferred Research LLC /ID# 227886, Miami, Florida
  - Neurology & Pain Medicine /ID# 240168, Miami, Florida
  - Medical Research Group of Central Florida /ID# 231632, Orange City, Florida
  - Clinical Associates of Orlando, LLC /ID# 272619, Orlando, Florida
  - Suncoast Clinical Research - Palm Harbor /ID# 229337, Palm Harbor, Florida
  - Asclepes Research Centers - Spring Hill /ID# 229815, Spring Hill, Florida
  - University of South Florida- Neuroscience Institute /ID# 229324, Tampa, Florida
  - Encore Medical Research - Weston /ID# 246809, Weston, Florida
  - Pediatric Neurology and Epilepsy Specialists /ID# 229967, Winter Park, Florida
  - Treken Primary Care /ID# 240586, Atlanta, Georgia
  - Rare Disease Research, LLC /ID# 231046, Atlanta, Georgia
  - Clinical Integrative Research Center of Atlanta (CIRCA) /ID# 231134, Atlanta, Georgia
  - Coastal Georgia Child Neurology /ID# 231409, Brunswick, Georgia
  - CenExcel iResearch LLC /ID# 227903, Decatur, Georgia
  - Velocity Clinical Research - Savannah. /ID# 228992, Savannah, Georgia
  - Sleep Care Research Institute d/b/a Clinical Research Institute /ID# 231738, Stockbridge, Georgia
  - Velocity Clinical Research - Boise /ID# 231871, Meridian, Idaho
  - Chicago Headache Center & Research Institute /ID# 248625, Chicago, Illinois
  - Ascension Saint Alexius /ID# 275261, Hoffman Estates, Illinois
  - Accellacare - McFarland Clinic /ID# 229789, Ames, Iowa
  - College Park Family Care Center Overland Park /ID# 231456, Overland Park, Kansas
  - Clinical Associates Midwest, LLC /ID# 274315, Overland Park, Kansas
  - Psychiatric Associates /ID# 230872, Overland Park, Kansas
  - Alliance for Multispecialty Research - Wichita East /ID# 234126, Wichita, Kansas
  - University of Kentucky Chandler Medical Center. /ID# 230827, Lexington, Kentucky
  - Pharmasite Research, Inc. /ID# 227908, Baltimore, Maryland
  - Minneapolis Clinic of Neurology - Burnsville /ID# 232551, Burnsville, Minnesota
  - MediSync Clinical Research Hattiesburg Clinic /ID# 233326, Petal, Mississippi
  - Proven Endpoints LLC /ID# 239513, Ridgeland, Mississippi
  - Sharlin Health and Neurology /ID# 229523, Ozark, Missouri
  - Cognitive Clinical Trials (CCT) - Papillion /ID# 232552, Papillion, Nebraska
  - Healthy Perspectives - Innovative Mental Health Services, PLLC /ID# 230312, Nashua, New Hampshire
  - Hunterdon Neurology /ID# 245648, Annandale, New Jersey
  - Goryeb Childrens Hospital /ID# 229507, Morristown, New Jersey
  - CVS HealthHUB - Runnemede /ID# 234233, Runnemede, New Jersey
  - Dent Neurologic Institute - Amherst /ID# 231182, Amherst, New York
  - Bioscience Research /ID# 232159, Mount Kisco, New York
  - Modern Migraine MD /ID# 258081, New York, New York
  - North Suffolk Neurology /ID# 230956, Port Jefferson Station, New York
  - SUNY Upstate Medical University /ID# 239898, Syracuse, New York
  - CVS HealthHUB - Charlotte /ID# 239530, Charlotte, North Carolina
  - OnSite Clinical Solutions, LLC - Hickory /ID# 227994, Hickory, North Carolina
  - Patient Priority Clinical Sites, LLC /ID# 238485, Cincinnati, Ohio
  - University Of Cincinnati Medical Center /ID# 231199, Cincinnati, Ohio
  - Cincinnati Childrens Hospital Medical Center /ID# 244689, Cincinnati, Ohio
  - Headache Center of Hope /ID# 242645, Cincinnati, Ohio
  - Centricity Research Columbus /ID# 231181, Columbus, Ohio
  - CincyScience /ID# 230046, West Chester, Ohio
  - IPS Research Company /ID# 227961, Oklahoma City, Oklahoma
  - Providence Brain and Spine Institute /ID# 231607, Portland, Oregon
  - Children's Hospital of Philadelphia - Main /ID# 232487, Philadelphia, Pennsylvania
  - Frontier Clinical Research, LLC - Scottdale /ID# 231913, Scottdale, Pennsylvania
  - Frontier Clinical Research - Smithfield /ID# 231912, Smithfield, Pennsylvania
  - Coastal Pediatric Research /ID# 238616, Charleston, South Carolina
  - Tribe Clinical Research LLC /ID# 230422, Greenville, South Carolina
  - Duplicate_Premier Neurology, P.C. /ID# 227999, Greer, South Carolina
  - Access Clinical Trials, Inc. /ID# 228002, Nashville, Tennessee
  - UT Health Austin at Dell Children's Neurology Clinic /ID# 244266, Austin, Texas
  - Austin Regional Clinic - ARC Four Points /ID# 276301, Austin, Texas
  - BioBehavioral Research of Austin /ID# 230529, Austin, Texas
  - Velocity Clinical Research, Austin /ID# 230557, Austin, Texas
  - Tekton Research - Beaumont /ID# 231207, Beaumont, Texas
  - Relaro Medical Trials /ID# 239642, Dallas, Texas
  - Cedar Health Research /ID# 228003, Dallas, Texas
  - Epic Medical Research - DeSoto /ID# 274314, DeSoto, Texas
  - 3A Research - East El Paso /ID# 239193, El Paso, Texas
  - Earle Research /ID# 231548, Friendswood, Texas
  - Innovare Research Group, LLC /ID# 277617, Friendswood, Texas
  - DM Clinical Research /ID# 229826, Houston, Texas
  - Houston Clinical Research Associates /ID# 244889, Houston, Texas
  - Pioneer Research Solutions - Houston - Stancliff Road /ID# 274316, Houston, Texas
  - Sante Clinical Research /ID# 246503, Kerrville, Texas
  - FMC Science /ID# 231915, Lampasas, Texas
  - Livingspring Family Medical Center /ID# 249869, Mansfield, Texas
  - AIM Trials /ID# 230142, Plano, Texas
  - Road Runner Research /ID# 230527, San Antonio, Texas
  - Family Psychiatry of The Woodlands /ID# 230163, The Woodlands, Texas
  - ClinPoint Trials /ID# 230295, Waxahachie, Texas
  - Pantheon Clinical Research /ID# 250703, Bountiful, Utah
  - Highland Clinical Research /ID# 239362, Salt Lake City, Utah
  - University of Utah Health Hospital /ID# 230908, Salt Lake City, Utah
  - Neuropsychiatric Associates LLC/DBA Woodstock Research Center /ID# 238976, Woodstock, Vermont
  - Office of Maria Ona /ID# 234232, Franklin, Virginia
  - Children's Hospital of The King's Daughters - Children's Medical Tower /ID# 230581, Norfolk, Virginia
  - National Clinical Research /ID# 231320, Richmond, Virginia
  - Core Clinical Research /ID# 227904, Everett, Washington
  - Frontier Clinical Research - Kingwood /ID# 231914, Kingwood, West Virginia
  - Mind+ Neurology /ID# 275529, Mequon, Wisconsin
- Puerto Rico (4):
  - Clinical Research Investigator Group, LLC /ID# 267454, Bayamón
  - Puerto Rico Health Institute /ID# 249162, Dorado
  - GCM Medical Group PSC /ID# 249643, San Juan
  - CMRC Headlands LLC /ID# 265301, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/